CLINICAL TRIAL: NCT07070050
Title: Continuous vs. Bolus Administration of NSAIDs After Laparoscopic Surgery for Multimodal Analgesia: Pilot Randomized Controlled Trial
Brief Title: Continuous vs. Bolus Administration of NSAIDs After Laparoscopic Surgery for Multimodal Analgesia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CALM
Record Dates: First submitted 2025-06-30; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Analgesic Drugs; Analgesic, Nonopioid; Analgesic Efficacy; Analgetic Consumption; Postoperative Care; Pain Management
Keywords: NSAID; pain management; analgesia; postoperative care; analgesic drug
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSAID bolus injection (Active Comparator)
  Interventions: Drug: Ibuprofen bolus injection
- NSAID continuous infusion (Experimental)
  Interventions: Drug: Ibuprofen continuous infusion

INTERVENTIONS:
Drug: Ibuprofen continuous infusion — 1. The first bolus: ibuprofen 400 mg diluted in 0,9% NaCl 200 ml is intravenous injected during the first hour right after the admission to the department. The drug is injected during the first hour at the rate of 4 mg/kg/h for the ideal body weight.
  2. Continuous infusion:
     * Ibuprofen 1200 mg diluted in 0,9% NaCl 300 ml is intravenous injected on the first day with the speed of 1 mg/kg/h (for the ideal body weight) during the remaining 23 hours.
     * On the second day the intravenous infusion of ibuprofen 1600 mg diluted in 0,9% NaCl 400 ml with the speed of 1 mg/kg/h is continued during the 24 hours.
  3. Imitation of bolus: Every 8 hours placebo (0, 9% NaCl 200 ml) is intravenous injected to create an imitation of bolus injection. Placebo is injected during the first hour.
  Arms: NSAID continuous infusion
Drug: Ibuprofen bolus injection — 1. The first bolus: ibuprofen 400 mg diluted in 0, 9% NaCl 200 ml is intravenous injected during the first hour right after the admission to the department. The drug is injected during the first hour at the rate of 4 mg/kg/h for the ideal body weight.
  2. Bolus injection:
     * Every 8 hours a intravenous bolus of ibuprofen 800 mg diluted in 0,9% NaCl 200 ml is injected during 1 hour (3 boluses per day in total).
     * On the second day the every 8 hours intravenous bolus of ibuprofen 800 mg diluted in 0, 9% NaCl 200 ml is injected during 1 hour (3 boluses per day in total).
  3. Placebo continuous infusion:
  Between the boluses a placebo (0,9% NaCl) continuous intravenous infusion is performed with the speed imitating the speed of ibuprofen infusion in the experimental group.
  Arms: NSAID bolus injection

SUMMARY:
Currently the prevalent approach to perioperative management of patients is ERAS (Enhanced Recovery After Surgery) concept. This approach includes numerous aspects, among which the perioperative use of multimodal analgesia takes one of the leading places. Within the ERAS guidelines all sorts of minimization of opioid analgesics use in schemes of postoperative analgesia are appreciated. Thus, new pharmacological approaches are being actively developed currently in order to achieve adequate analgesia and to minimize the use of this group of drugs.

One of the most perspective trends within the multimodal analgesia concept is continuous infusion of non-steroidal anti-inflammatory drugs (NSAID). Up to date there are papers that both confirm the effectiveness of this method for maintaining adequate postoperative analgesia and show its limitations and deny the advantages of the continuous use of NSAID.

Up to this time the main attention of the medical community was paid for such drugs as paracetamol and ketoprofen. Nevertheless, one of the most common and safe NSAID is ibuprofen. In spite of this, there are no studies that explore the effectiveness of the continuous infusion of this drug. Thus, the lack of even low-quality evidence led to setting up a study of effectiveness and safety of continuous infusion of ibuprofen in comparison to its bolus injection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Elective laparoscopic surgery
* General anesthesia
* Signed informed consent from the patient to participate in the study
* RASS scale from -2 to +1 on admission to a surgical department or ICU

Exclusion Criteria:

* History of ibuprofen allergy
* Active erosive or ulcerative lesions of the gastrointestinal tract
* Chronic use of opioid analgesics or NSAIDs prior to enrollment
* Chronic kidney disease ≥ 3b stage according to the KDIGO classification
* Liver dysfunction (three times exceeding the upper reference limit of ALT or AST)
* A history of bronchial asthma
* A history of hereditary coagulopathies
* A history of use of anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | up to 28 days
  Evaluation of the overall consumption of opioid analgesics after surgery during the whole postoperative period

SECONDARY OUTCOMES:
Pain intensity assessment | From admission to ICU until 48 hours postoperatively
  Evaluation of postoperative pain intensity using the Numerical Rating Scale (NRS); measurements at regular intervals and before rescue analgesia if pain exceeds NRS >5. The maximum value is 10, the minimum value is 0. The higher the value, the more severe patient's pain (worse).

OTHER OUTCOMES:
NSAID-related Adverse Effects | up to 28 days
  Incidence and severity of adverse effects including respiratory depression, gastrointestinal dysfunction, hepatotoxicity, renal dysfunction, allergic reactions, and CNS effects.
Length of ICU stay | 1 year
  The number of days between the day of discharge from the ICU (or in-hospital death) after initial admission and the day of randomization.
Length of Hospital Stay | 1 year
  The number of days between the day of discharge from the hospital (or in-hospital death) after initial admission and the day of randomization.
ICU Readmission | Within 28 days from randomization
  Incidence of readmission to the intensive care unit within 28 days from the day of randomization.
In-hospital mortality | 1 year
  Number of patients who die from any cause during initial hospitalization
28-days mortality | From randomization to 28 days
  Number of patients who die from any cause within28 days after randomization
6-month mortality | From randomization to 6 months
  Number of patients who die from any cause within 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Valery Likhvantsev, PhD, Principal Investigator — Federal Research and Clinical Center of Intensive Care Medicine and Rehabilitology
Locations (1):
- City Clinical Hospital named after S.S. Yudin, Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: No